CLINICAL TRIAL: NCT05304637
Title: Usability, Immediate, and 30 Day Effect of External Neuromodulation With iTEAR100 Generation 2 in Dry Eye Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olympic Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-011
Record Dates: First submitted 2022-03-09; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Open labe therapeutic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Therapy Arm (Experimental): Patient receive iTEAR100 treatment
  Interventions: Device: iTEAR100 treatment

INTERVENTIONS:
Device: iTEAR100 treatment — Vibratory energy to the external nasal nerve

SUMMARY:
iTEAR generation 2 will be supplied t eligible subjects at Day 0. At Day 30, symptom questionnaires and ophthalmic exam will be performed.

DETAILED DESCRIPTION:
TEAR generation 2 will be supplied t eligible subjects at Day 0. At Day 30, symptom questionnaires and ophthalmic exam will be performed. At both exam days, a Schirmer test before and after will be performed as well as parameters which indicate immediate effect of treatment and treatment over the 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Dry eye

Exclusion Criteria:

* unable to read consent
* investigator discretion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Schirmer score | within 5 minutes of stimulation
  Difference between Schirmer score measured before stimulation and after stimulation at each visit

SECONDARY OUTCOMES:
Symptom Scores | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Olympic Ophthalmics, Issaquah, Washington
  - Periman Eye Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No